CLINICAL TRIAL: NCT03829579
Title: Esketamine Single Patient Request
Brief Title: Pre-Approval Access to Esketamine Nasal Spray for the Treatment of Treatment-Resistant Depression (TRD)
Status: Approved for marketing | Type: Expanded Access
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108572; 54135419TRD3012 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-02-01; First posted 2019-02-04 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Depressive Disorder, Treatment-Resistant
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Esketamine

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Esketamine — Participants will self-administer esketamine nasal spray, under the supervision of the healthcare professional at the site of care. A starting dose of 56 milligram (mg) will be administered intranasally into each nostril on Day 1 with subsequent doses of 56 mg or 84 mg administered during Weeks 1-4 (2 treatment sessions per week). For participants who respond, treatment is continued as follows: 56 mg or 84 mg of esketamine nasal spray during Weeks 5-8 (once weekly), and Week 9 onwards (every 2 weeks or once weekly), with period re-evaluation to determine the need for continued treatment. Doses will be adjusted based on efficacy and tolerability to the previous dosing.

SUMMARY:
This is a pre-approval access program (PAAP) for eligible participants. The main purpose of this program is to provide access to esketamine nasal spray to eligible participant with treatment-resistant depression (TRD), who have exhausted all other treatment options, including all alternative treatment options with marketed therapies.

ELIGIBILITY:
Inclusion Criteria:

* Must have an unmet medical need to treat treatment-resistant depression (TRD) with esketamine nasal spray, an investigational compound, that has not been approved by any health authority. This means no other treatment options are available and the participant must be unable to participate in a clinical trial; for example, because they do not fulfill the eligibility criteria of the protocol or there are no trial sites within a reasonable distance of where they reside
* Must not participate in a clinical trial or be concurrently treated with an investigational drug when being treated with esketamine nasal spray
* Participants must have TRD with the diagnosis verified by a psychiatrist, and have exhausted all other options including all alternative treatment options with marketed therapies, specifically:

  1. Participant must meet the Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 diagnostic criteria for single-episode major depressive episode (major depressive disorder [MDD]) (if single-episode MDD, the duration must be greater than [>]2 years) or recurrent MDD, without psychotic features.
  2. Participant must have had nonresponse to 2 or more oral antidepressant treatments in the current episode of depression confirmed by documented medical history and/or pharmacy/prescription records to meet criteria for TRD and have failed at least one augmentation strategy (for example, atypical antipsychotics such as aripiprazole or quetiapine, lithium, thyroid hormones, bupropion, etc) and have failed an adequate course (greater than or equal to [>=] 7 unilateral [UL] sessions) of, or have a contraindication to electro-convulsive therapy (ECT) and transcranial magnetic stimulation (TMS)
* Participants must have exhausted clinical trials, early access programs or named patient programs that may be available in their region
* Participants must have moderate to severe depression per clinical judgment

Exclusion Criteria:

* The participant's depressive symptoms have previously demonstrated nonresponse to Esketamine Nasal Spray or ketamine in the current major depressive episode per clinical judgment
* Participant has a current or prior DSM-5 diagnosis of a psychotic disorder or MDD with psychosis, bipolar or related disorders, comorbid obsessive- compulsive disorder, intellectual disability (only DSM-5 diagnostic code 319), borderline personality disorder, antisocial personality disorder, histrionic personality disorder, or narcissistic personality disorder
* Participant has homicidal ideation/intent or has suicidal ideation with some intent to act within 6 months or a history of suicidal behavior within the past year, per the requesting psychiatrist's clinical judgment
* Participant has a history of moderate or severe substance or alcohol use disorder according to DSM-5 criteria, except nicotine or caffeine, within 6 months before the start of the first dose.

  a) A history (lifetime) of ketamine, phencyclidine (PCP), lysergic acid diethylamide (LSD), or 3, 4-methylenedioxy-methamphetamine (MDMA) hallucinogen-related use disorder is exclusionary
* Participants with a current or past history of seizures (uncomplicated childhood febrile seizures with no sequelae are not exclusionary)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC